CLINICAL TRIAL: NCT00663754
Title: Eating Disorder Prevention Program Effectiveness Trial
Brief Title: Effectiveness of a Dissonance-Based Eating Disorder Prevention Program (The Body Project II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH070699 (NIH); R01MH070699 (NIH); DSIR 84-CTP
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Eating Disorders
Keywords: Body Image
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Participants will receive a mailed brochure about body image only.
  Interventions: Behavioral: Educational brochure
- 2 (Active Comparator): Participants will receive the 4-hour dissonance-based eating disorder prevention program.
  Interventions: Behavioral: Dissonance-based eating disorder prevention program
- 3 (Experimental): Participants will receive the 8-hour dissonance-based eating disorder prevention program.
  Interventions: Behavioral: Dissonance-based eating disorder prevention program

INTERVENTIONS:
Behavioral: Dissonance-based eating disorder prevention program — Participants will engage in verbal, written, and behavioral exercises in which they will critique the thin ideal. These exercises will be conducted in sessions and in homework activities. The exercises will aim to increase body image satisfaction by helping participants to think critically about the thin ideal and to discuss some of the problems associated with the pursuit of this ideal.
  Arms: 2; 3
Behavioral: Educational brochure — Participants will receive a mailed educational brochure about a healthy body image only.
  Arms: 1

SUMMARY:
This study will evaluate the effectiveness of dissonance-based eating disorder prevention programs in reducing body dissatisfaction among young women with body image concerns.

DETAILED DESCRIPTION:
It is estimated that up to 80% of young adult women in the United States are dissatisfied with their appearance, particularly their weight. Young women's perception of the ideal body type is influenced by many factors, including peers, parents, and the media. Body dissatisfaction is associated with an increased risk of depression and eating disorders, making programs to reduce body image issues in young women important. Programs that target eating disorder prevention through promoting healthy behaviors and critiquing the thin ideal may be an effective means of increasing body satisfaction among young women. Particularly, a dissonance-based eating disorder prevention program that assesses the thin ideal through verbal, written, and behavioral exercises may be the best means of addressing body image concerns. This study will evaluate the effectiveness of dissonance-based eating disorder prevention programs in reducing body dissatisfaction among young women with body image concerns.

Participation in this study will last 2 years and will involve both parent and daughter participants. Study participation for parent participants will include three 15-minute interviews conducted at baseline and Years 1 and 2. The interviews will focus on their daughters' social adjustment, performance in school, relationships with others, hobbies, and related topics. Daughter participants will still be allowed to partake in the study even if their parents do not complete all three interviews.

All potential daughter participants will first complete a 20-minute interview regarding their eating habits and mental health. Eligible participants will then be assigned to one of three programs designed to improve body image satisfaction:

* Program 1 will consist of the distribution of an educational brochure about a healthy body image.
* Program 2 will involve four 1-hour meetings during which participants will complete a series of verbal and written exercises. The exercises will aim to increase body image satisfaction by helping participants to think critically about the thin ideal and to discuss some of the problems associated with the pursuit of this ideal.
* Program 3 will include eight 1-hour meetings during which participants will also complete a series of verbal and written exercises. The exercises will aim to increase body image satisfaction by helping participants to think critically about the thin ideal and by promoting healthy eating and exercise habits.

Participants in all programs will complete brief surveys and interviews about their attitudes and behaviors at baseline, at treatment completion, and at three other points during the 2 years from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported body image concerns

Exclusion Criteria:

* Meets diagnostic and statistical manual (DSM-IV) criteria for anorexia nervosa, bulimia nervosa, or binge eating disorder

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 306 (Actual)
Dates: Start 2005-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Diagnostic Interview | Measured at baseline, post-treatment, Month 6, and Years 1 and 2

SECONDARY OUTCOMES:
Ideal-Body Stereotype Scale-Revised, Satisfaction and Dissatisfaction with Body Parts Scale, Dutch Restrained Eating Scale, Positive Affect and Negative Affect Scale-Revised, and Beliefs About Appearance Scale | Measured at baseline, post-treatment, Month 6, and Years 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, Principal Investigator — Oregon Research Institute; Paul Rhode, Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

REFERENCES:
- [Derived] Stice E, Desjardins C, Shaw H, Siegel S, Gee K, Rohde P. Prevalence, incidence, impairment, course, and diagnostic progression and transition of eating disorders, overweight, and obesity in a large prospective study of high-risk young women. J Psychopathol Clin Sci. 2025 May;134(4):427-437. doi: 10.1037/abn0000965. Epub 2024 Nov 7. PMID 39509183
- [Derived] Stice E, Desjardins CD, Rohde P. Young women who develop anorexia nervosa exhibit a persistently low premorbid body weight on average: A longitudinal investigation of an important etiologic clue. J Psychopathol Clin Sci. 2022 Jul;131(5):479-492. doi: 10.1037/abn0000762. Epub 2022 Jun 2. PMID 35653756
- [Derived] Stice E, Desjardins CD, Rohde P, Shaw H. Sequencing of symptom emergence in anorexia nervosa, bulimia nervosa, binge eating disorder, and purging disorder and relations of prodromal symptoms to future onset of these disorders. J Abnorm Psychol. 2021 May;130(4):377-387. doi: 10.1037/abn0000666. PMID 34180702